CLINICAL TRIAL: NCT06436586
Title: Impact of HLA Evolutionary Divergence and HLA Donor-recipient Molecular Mismatches on Kidney Allograft Rejection: a Population-based Study
Brief Title: Impact of HLA Evolutionary Divergence and HLA Donor-recipient Molecular Mismatches on Kidney Allograft Rejection
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: HLA_kidney_001
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The Human Leucocyte Antigen (HLA) system is pivotal in kidney transplant rejection. In-silico methods such as HLA eplet mismatches and PIRCHE-II scores have emerged to refine HLA immunogenicity assessment and stratify patients for immunological risk. However, large-scale studies in unselected large kidney transplant cohorts are lacking to support their broader clinical applicability. Additionally, recent studies on HLA evolutionary divergence (HED), quantifying HLA polymorphism, highlight its potential impact on rejection. Yet, the association of HED with kidney allograft rejection or de novo DSA occurrence remains unexplored in kidney transplantation.

The complexity introduced by diverse in-silico methods for assessing HLA immunogenicity necessitates further research to comprehensively understand their role in relation to kidney allograft rejection.

This project thus aims to investigate the association between various aspects of HLA immunogenicity, including HLA molecular mismatches and HLA evolutionary divergence, along with standard immunological and clinical parameters assessed at the time of transplantation, with the occurrence of antibody-mediated rejection and de novo DSA formation post-transplant in a large, comprehensively annotated kidney transplant cohort.

ELIGIBILITY:
Inclusion Criteria:

* Living or deceased donor kidney recipient transplanted after 2004
* Kidney recipient older than 18 years of age
* Written informed consent at the time of transplantation for the center database

Exclusion Criteria:

* Combined transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients from four French referral centers
Sampling Method: Non-Probability Sample
Enrollment: 5159 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Antibody-mediated rejection | from 02/01/2004 to 25/01/2021

SECONDARY OUTCOMES:
De novo anti-HLA donor-specific antibody | from 02/01/2004 to 25/01/2021

CONTACTS AND LOCATIONS:
Locations (1):
- Paris Translational Research Center for Organ Transplantation, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bestard O, Thaunat O, Bellini MI, Bohmig GA, Budde K, Claas F, Couzi L, Furian L, Heemann U, Mamode N, Oberbauer R, Pengel L, Schneeberger S, Naesens M. Alloimmune Risk Stratification for Kidney Transplant Rejection. Transpl Int. 2022 May 20;35:10138. doi: 10.3389/ti.2022.10138. eCollection 2022. PMID 35669972
- [Background] Sellares J, de Freitas DG, Mengel M, Reeve J, Einecke G, Sis B, Hidalgo LG, Famulski K, Matas A, Halloran PF. Understanding the causes of kidney transplant failure: the dominant role of antibody-mediated rejection and nonadherence. Am J Transplant. 2012 Feb;12(2):388-99. doi: 10.1111/j.1600-6143.2011.03840.x. Epub 2011 Nov 14. PMID 22081892
- [Background] Wiebe C, Rush DN, Nevins TE, Birk PE, Blydt-Hansen T, Gibson IW, Goldberg A, Ho J, Karpinski M, Pochinco D, Sharma A, Storsley L, Matas AJ, Nickerson PW. Class II Eplet Mismatch Modulates Tacrolimus Trough Levels Required to Prevent Donor-Specific Antibody Development. J Am Soc Nephrol. 2017 Nov;28(11):3353-3362. doi: 10.1681/ASN.2017030287. Epub 2017 Jul 20. PMID 28729289
- [Background] Lachmann N, Niemann M, Reinke P, Budde K, Schmidt D, Halleck F, Pruss A, Schonemann C, Spierings E, Staeck O. Donor-Recipient Matching Based on Predicted Indirectly Recognizable HLA Epitopes Independently Predicts the Incidence of De Novo Donor-Specific HLA Antibodies Following Renal Transplantation. Am J Transplant. 2017 Dec;17(12):3076-3086. doi: 10.1111/ajt.14393. Epub 2017 Jul 28. PMID 28613392
- [Background] Feray C, Taupin JL, Sebagh M, Allain V, Demir Z, Allard MA, Desterke C, Coilly A, Saliba F, Vibert E, Azoulay D, Guettier C, Chatton A, Debray D, Caillat-Zucman S, Samuel D. Donor HLA Class 1 Evolutionary Divergence Is a Major Predictor of Liver Allograft Rejection : A Retrospective Cohort Study. Ann Intern Med. 2021 Oct;174(10):1385-1394. doi: 10.7326/M20-7957. Epub 2021 Aug 24. PMID 34424731
- [Derived] Demir Z, Raynaud M, Divard G, Louis K, Truchot A, Niemann M, Ponsirenas R, Aubert O, Del Bello A, Hertig A, Anglicheau D, Dale B, Kamar N, Mangiola M, Zeevi A, Lefaucheur C, Loupy A. Impact of HLA evolutionary divergence and donor-recipient molecular mismatches on antibody-mediated rejection of kidney allografts. Nat Commun. 2025 Jul 1;16(1):5692. doi: 10.1038/s41467-025-60485-y. PMID 40592858